CLINICAL TRIAL: NCT07149272
Title: Lactate Kinetics Analysis Related to Low-Intensity Resistance Exercise: Randomized Control Trial
Brief Title: Lactate Kinetics Analysis Related to Low-Intensity Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Melinda Harini, Dr. dr. Melinda Harini, Sp.K.F.R., Ger. (K), Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET-261/UN2.F1/ETIK/PPM.00.02/
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Fatigue; Lactate
Keywords: Exercise; Geriatric; Lactate; Virtual Reality
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study utilized a two-arm, parallel-group, randomized controlled trial (RCT) design with single-blinding to evaluate the efficacy of Virtual Reality Exercise (VRE) as an adjuvant therapy for hospitalized geriatric patients. Sixty participants were randomly assigned to either a control group receiving conventional multimodal exercise or an intervention group receiving conventional exercise plus VRE using VRAGMENT software on Oculus Quest 2. Both groups underwent simultaneous interventions with outcomes measured at baseline and one week post-intervention, focusing on lactate kinetics as the primary outcome. The single-blind design ensured participants were unaware of their group allocation to minimize bias, while clinicians administering the interventions remained unblinded due to the nature of the VR therapy.
Who Masked: Participant
Masking Description: Participants were blinded to group allocation (control vs. VRE intervention) to minimize performance bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Conventional multimodal exercise (standard care)
- VRE Intervention Group (Experimental): Conventional exercise + Virtual Reality Exercise (VRAGMENT software on Oculus Quest 2)
  Interventions: Device: Virtual Reality Exercise (VRE) using VRAGMENT software

INTERVENTIONS:
Device: Virtual Reality Exercise (VRE) using VRAGMENT software — Adjuvant Virtual Reality Exercise (VRE) delivered via Oculus Quest 2 headset with VRAGMENT software, a culturally adapted VR program simulating daily activities (e.g., grocery shopping, phone calls) to induce physical movement. Participants received VRE alongside conventional multimodal exercise (breathing, resistance, aerobic) during hospitalization. Sessions were tailored to individual clinical conditions and aimed to improve fatigue and mobility through gamified rehabilitation
  Other Names: VRAGMENT
  Arms: VRE Intervention Group

SUMMARY:
The goal of this study aims to analyze lactate kinetics as an exercise response after conventional multimodal exercise and virtual reality exercise (VRE) in hospitalized geriatric. The main question it aims to answer are:

1. are there any difference in post exercise lactate at day 1 and 7 between the two groups?
2. does the lactate concentration reduces after low intensity resistance exercise in subject with high resting lactate?

Participants were randomized into control and VRE group. Peripheral blood lactate was taken immediately before and after low-intensity resistance exercise at baseline and one week after

DETAILED DESCRIPTION:
Sixty geriatric patients were recruited during their hospitalization at RSUPN Dr. Cipto Mangunkusumo (RSCM). Subjects were randomized into control and intervention group. Both groups get conventional multimodal exercise, the intervention group gets additional VRE as adjuvant therapy. Exercise prescription was given after the subjects going through functional assessment conducted by physiatrists. The prescription described the frequency, intensity, interval, and type of exercise that is adjusted to subject's clinical condition. Each subject could have more than one type of exercise, but the most common combination consists of breathing, resistance, and aerobic exercises. VRAGMENT software was administered as VRE to the intervention group. In VRAGMENT, subjects should make phone call, groceries and making payment. Those activities in virtual environment initiated real movement of neck, trunk, arms, and legs. Capillary blood lactate sample was examined using StatStrip® from Nova Biomedical. Measurement range of StatStrip® is 0,3 - 20,0 mmol/L. Lactate examination conducts at baseline and one week after the exercise program. Blood samples were collected immediately pre and post-standardized low-intensity resistance training. The data collected were analyzed using SPSS statistics (version 24.0).

ELIGIBILITY:
Inclusion Criteria:

* Patient age 60-90 years old in acute geriatric ward
* mobilization level 3 and 4
* able to communicate and follow instructions

Exclusion Criteria:

* VR Sickness
* severe psychosocial problems
* severe caregiver burden

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Post-Exercise Blood Lactate Concentration (mmol/L) | The change from pre- to post-exercise is measured on Day 1 and again on Day 7. The outcome is the comparison of these changes between the two days
  The absolute change in capillary blood lactate concentration (mmol/L) from pre-exercise to immediately post-exercise. This change will be calculated at two time points: at baseline (Day 1) and one week post-intervention (Day 7). The difference between the Day 7 change and the Day 1 change will be the primary outcome. Measurements will be taken using the StatStrip® Lactate Meter

SECONDARY OUTCOMES:
Lactate Clearance Rate (% change per minute) | Measured during the recovery phase on Day 1 and Day 7. The outcome is the comparison of the clearance rates between the two days
  The rate at which blood lactate is cleared following exercise, calculated as the percentage decrease in lactate concentration from the immediate post-exercise peak to a subsequent measurement. This provides a kinetic measure of metabolic recovery
Qualitative Pattern of Fatigue via Lactate Kinetics | Patterns are assessed by comparing the kinetic profiles from Day 1 to Day 7
  A qualitative assessment of the overall lactate kinetic response (combining the post-exercise change and clearance rate) to infer clinical patterns of fatigue improvement

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality

REFERENCES:
- [Background] Cortes-Perez I, Sanchez-Alcala M, Nieto-Escamez FA, Castellote-Caballero Y, Obrero-Gaitan E, Osuna-Perez MC. Virtual Reality-Based Therapy Improves Fatigue, Impact, and Quality of Life in Patients with Multiple Sclerosis. A Systematic Review with a Meta-Analysis. Sensors (Basel). 2021 Nov 6;21(21):7389. doi: 10.3390/s21217389. PMID 34770694
- [Background] Vavricka J, Broz P, Follprecht D, Novak J, Krouzecky A. Modern Perspective of Lactate Metabolism. Physiol Res. 2024 Aug 31;73(4):499-514. doi: 10.33549/physiolres.935331. PMID 39264074
- [Background] Goodwin ML, Harris JE, Hernandez A, Gladden LB. Blood lactate measurements and analysis during exercise: a guide for clinicians. J Diabetes Sci Technol. 2007 Jul;1(4):558-69. doi: 10.1177/193229680700100414. PMID 19885119
- [Background] Cho H, Sohng KY. The effect of a virtual reality exercise program on physical fitness, body composition, and fatigue in hemodialysis patients. J Phys Ther Sci. 2014 Oct;26(10):1661-5. doi: 10.1589/jpts.26.1661. Epub 2014 Oct 28. PMID 25364137
- [Background] Schneider SM, Hood LE. Virtual reality: a distraction intervention for chemotherapy. Oncol Nurs Forum. 2007 Jan;34(1):39-46. doi: 10.1188/07.ONF.39-46. PMID 17562631
- [Background] Patino-Hernandez D, David-Pardo DG, Borda MG, Perez-Zepeda MU, Cano-Gutierrez C. Association of Fatigue With Sarcopenia and its Elements: A Secondary Analysis of SABE-Bogota. Gerontol Geriatr Med. 2017 Apr 10;3:2333721417703734. doi: 10.1177/2333721417703734. eCollection 2017 Jan-Dec. PMID 28474000
- [Background] Ioannou A, Papastavrou E, Avraamides MN, Charalambous A. Virtual Reality and Symptoms Management of Anxiety, Depression, Fatigue, and Pain: A Systematic Review. SAGE Open Nurs. 2020 Aug 27;6:2377960820936163. doi: 10.1177/2377960820936163. eCollection 2020 Jan-Dec. PMID 33415290

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT07149272/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT07149272/ICF_001.pdf